CLINICAL TRIAL: NCT04709081
Title: A Two-Part Phase 1 Study to Evaluate the Potential Drug Interaction Between ACH-0145228 and Midazolam, Digoxin, and Itraconazole in Healthy Adult Subjects
Brief Title: A Drug Interaction Study of ACH-0145228
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry); Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH228-003; CA28776 (Other: Celerion)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; Capsule; Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — Midazolam; Digoxin; Itraconazole

STUDY DESIGN:
Intervention Model Description: Part 1 and Part 2 could be conducted concurrently or separately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: ACH-0145228, Midazolam, and Digoxin (Experimental): Period 1: Participants received single doses of midazolam and digoxin.
  Period 2: Participants received ACH-0145228 twice daily, in addition to coadministration with single doses of midazolam and digoxin.
  Scheduled pharmacokinetics (PK) blood and urine samples were collected, with a washout period of at least 7 days between collection of the last PK blood sample in Period 1 and the first dose of ACH-0145228 in Period 2.
  Interventions: Drug: ACH-0145228; Drug: Midazolam; Drug: Digoxin
- Part 2: ACH-0145228 and Itraconazole (Experimental): Period 1: Participants received a single dose of ACH-0145228.
  Period 2: Participants received itraconazole once daily, in addition to coadministration with a single dose of ACH-0145228.
  Scheduled PK blood samples were collected, with a washout period of at least 2 days between collection of the last PK blood sample in Period 1 and the first dose of itraconazole in Period 2.
  Interventions: Drug: ACH-0145228; Drug: Itraconazole

INTERVENTIONS:
Drug: ACH-0145228 — ACH-0145228 was dosed as 2 x 60 milligram (mg) (Part 1) or 1 x 40 mg (Part 2) powder in capsules.
  Other Names: ALXN2050
Drug: Midazolam — Midazolam was dosed at 2 mg (1 milliliter [mL] of a 2 mg/mL syrup).
  Other Names: Midazolam HCl
  Arms: Part 1: ACH-0145228, Midazolam, and Digoxin
Drug: Digoxin — Digoxin was dosed as Lanoxin (or generic equivalent) at 1 x 0.25 mg tablet.
  Other Names: Lanoxin
  Arms: Part 1: ACH-0145228, Midazolam, and Digoxin
Drug: Itraconazole — Itraconazole was dosed as Sporanox (or generic equivalent) at 200 mg (20 mL of a 10 mg/mL oral solution).
  Other Names: Sporanox
  Arms: Part 2: ACH-0145228 and Itraconazole

SUMMARY:
This was a 2-part study (Part 1 and Part 2), with each part being an open-label, fixed sequence, 2-period study in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
2. No clinically significant history or presence of electrocardiogram abnormalities at screening and prior to first dosing in Period 1.
3. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.
4. Female participants must be of non-childbearing potential and need not employ a method of contraception.

Exclusion Criteria:

1. Clinically significant laboratory abnormalities.
2. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
3. History or presence of drug or alcohol abuse within previous 2 years, current tobacco/nicotine user, or positive for alcohol and/or drug screen at screening or Day -1 of Period 1.
4. History or presence of clinically significant seizures, head injury, or head trauma.
5. History of procedures that could alter absorption or excretion of orally administered drugs.
6. A history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
7. Body temperature ≥ 38.0°Celsius at screening or prior to first dosing in Period 1.
8. Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing, or receipt of blood products within 6 months prior to first dosing.
9. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever is longer.
10. History or presence of any risk factors for Torsades de Pointes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-12-22 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Part 1: Area Under The Concentration Versus Time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Single-dose Midazolam Under Multiple Doses Of ACH-0145228 | Up to 24 hours postdose
Part 1: Maximum Observed Concentration (Cmax) Of Single-dose Midazolam Under Multiple Doses Of ACH-0145228 | Up to 24 hours postdose
Part 1: Time To Maximum Observed Concentration (Tmax) Of Single-dose Midazolam Under Multiple Doses Of ACH-0145228 | Up to 24 hours postdose
Part 1: AUC0-inf Of Single-dose Digoxin Under Multiple Doses Of ACH-0145228 | Up to 168 hours postdose
Part 1: Cmax Of Single-dose Digoxin Under Multiple Doses Of ACH-0145228 | Up to 168 hours postdose
Part 1: Tmax Of Single-dose Digoxin Under Multiple Doses Of ACH-0145228 | Up to 168 hours postdose
Part 2: AUC0-inf Of Single-dose ACH-0145228 Under Multiple Doses Of Itraconazole | Up to 96 hours postdose
Part 2: Cmax Of Single-dose ACH-0145228 Under Multiple Doses Of Itraconazole | Up to 96 hours postdose
Part 2: Tmax Of Single-dose ACH-0145228 Under Multiple Doses Of Itraconazole | Up to 96 hours postdose

SECONDARY OUTCOMES:
Part 1: Number Of Participants With Treatment-emergent Adverse Events (TEAEs) After Multiple Doses Of ACH-0145228 Coadministered With A Single Dose Of Midazolam | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)
Part 1: Number Of Participants With TEAEs After Multiple Doses Of ACH-0145228 Coadministered With A Single Dose Of Digoxin | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)
Part 2: Number Of Participants With TEAEs After A Single Dose Of ACH-0145228 Coadministered With Multiple Doses Of Itraconazole | Day 1 (postdose) through follow-up (14 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No